CLINICAL TRIAL: NCT06343792
Title: Phase 2 Open Label Prospective Dose-Ranging Clinical Trial With Escalation and Expansion Cohorts to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Dosing, and Efficacy of RLS-0071 for the Treatment of Hospitalized Patients With Steroid-Refractory Acute Graft-versus-Host Disease
Brief Title: Safety, PK, PD, Dosing, and Efficacy of RLS-0071for the Treatment of Hospitalized Patients With Steroid-Refractory Acute Graft-versus-Host Disease
Acronym: AURORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ReAlta Life Sciences, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RLS-0071-203
Record Dates: First submitted 2024-03-14; First posted 2024-04-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Steroid Refractory GVHD
MeSH Terms: interventions — RLS-0071

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- RLS-0071Cohort 1 (Experimental): 10 mg/kg Q8H RLS-0071 for 7 days
  Interventions: Drug: RLS-0071
- RLS-0071 Cohort 2 (Experimental): 10 mg/kg Q8H RLS-0071 for 14 days with concurrent ruxolitinib
  Interventions: Drug: RLS-0071
- RLS-0071 Cohort 3 (Experimental): 20 mg/kg Q8H RLS-0071 for 14 days with concurrent ruxolitinib
  Interventions: Drug: RLS-0071
- RLS-0071 Cohort 4 (Experimental): 10 mg/kg Q8H RLS-0071 for 7 days and then 10 mg/kg QD RLS-0071 for 7 days with concurrent ruxolitinib
  Interventions: Drug: RLS-0071
- RLS-0071 Cohort 5 (Experimental): 20 mg/kg Q8H RLS-0071 for 7 days and then 20 mg/kg QD RLS-0071 for 7 days with concurrent ruxolitinib
  Interventions: Drug: RLS-0071
- RLS-0071 Expansion Cohort 1 (Experimental): 12 participants will receive 10 mg/kg Q8H RLS-0071 for 14 days
  Interventions: Drug: RLS-0071
- RLS-0071 Expansion Cohort 2 (Experimental): 12 participants will receive 20 mg/kg Q8H RLS-0071 for 14 days
  Interventions: Drug: RLS-0071

INTERVENTIONS:
Drug: RLS-0071 — RLS-0071 will be administered for 7 or 14 days according to the assigned dose group.

SUMMARY:
This study is a Open Label Prospective Dose-Ranging Escalation and Expansion Trial to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Dosing, and Efficacy of RLS-0071 for the secondary treatment of acute Graft-versus-Host Disease (aGvHD) in hospitalized patients who are steroid-refractory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults or adolescents (>12 years old).
* Hospitalized with steroid-refractory aGvHD (grade II-IV) after allo-HSCT
* Anticipated hospital length-of-stay of at least 1 week from the time of RLS-0071 initiation.
* No plans to add additional GvHD treatment medications or to add, dose-adjust, or discontinue GvHD prophylactic medications during the 7-days of RLS-0071 treatment.
* Neutrophil recovery following the stem-cell transplantation, defined as blood neutrophil count >500/mL for at least 3 consecutive measurements and not supported by growth factor supplementation
* Weight ≥40 kg and ≤ 140 kg at screening.

Exclusion Criteria:

* Has received more than 1 allo-HSCT
* Current, previous, or planned use of any systemic treatment in addition to or other than corticosteroids or ruxolitinib for aGvHD
* Previous failure of ruxolitinib treatment
* Uncontrolled GI infection
* Endoscopic and biopsy testing (if performed) that definitively rules out lower GI aGvHD
* Chronic GvHD
* Participants with evidence of relapsed primary disease, or participants who have been treated for relapse after the allo-HSCT was performed.
* Unresolved toxicity or complications (other than aGvHD) due to the allo-HSCT
* Any corticosteroid therapy for indications other than aGvHD at doses of methylprednisolone or equivalent >1 mg/kg per day within 7 days of enrollment.
* Severe organ dysfunction unrelated to underlying aGvHD
* Known hypersensitivity, allergy, or anaphylactic reaction to polyethylene glycol (PEG)
* Significant liver disease that is unrelated to GvHD
* Severe kidney disease
* Currently breast feeding.
* Known pregnancy, a positive pregnancy test at screening, or lactation for WOCBP.
* Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or human immunodeficiency virus (HIV)-1 or HIV-2.
* Active sepsis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Day 1 to Day 180
Overall Response Rate (ORR) of RLS-0071 | Day 1 to Day 28

SECONDARY OUTCOMES:
Incidence of refractoriness (to RLS-0071 +/- ruxolitinib) | Days 7, 14, 28, 56, and 180
Overall corticosteroid use | Days 7, 14, 28, 56, and 180
Initiation of additional or alternative treatment(s) for aGvHD (including an increase in steroid dose to >2 mg/kg methylprednisolone equivalent) | Day 1 - Day 180
Change or shift in Stage for lower GI aGvHD, liver aGvHD, skin aGvHD, or upper GI aGvHD from baseline based on MAGIC Criteria | Days 7, 14, 28, 56, and 180
Attainment of Stage 0 or 1 lower GI aGvHD, liver aGvHD, skin aGvHD, or upper GI aGvHD | Days 7, 14, 28, 56, and 180
Change or shift in overall Grade of aGvHD | Day 0 - Days 7, 14, 28, 56, and 180.
Overall survival | Day 1 - Day 180
Non-relapse mortality | Day 1 - Day 180
Duration of hospital stay | Day 1 - Day 180

CONTACTS AND LOCATIONS:
Locations (11):
- United States (6):
  - Site 1091, Duarte, California
  - Site 1343, Los Angeles, California
  - Site 1318, Atlanta, Georgia
  - Site 1068, St Louis, Missouri
  - Site 1100, Cincinnati, Ohio
  - Site 1382, Columbus, Ohio
- Site 3242, Freiburg im Breisgau, Germany
- Spain (4):
  - Site 3101, Seville, SE
  - Site 3360, Madrid
  - Site 3227, Salamanca
  - Site 3101, Seville